CLINICAL TRIAL: NCT04719403
Title: Determining the Feasibility, Acceptability, and Potential Effectiveness of Sharing Video Recordings of Multidisciplinary ALS Clinics With Patients and Their Caregivers
Brief Title: Determining Feasibility and Acceptability of Sharing Video Recordings With Patients With ALS and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: The Diamond Endowment Project (Unknown)
Responsible Party: Principal Investigator, Paul J. Barr, Associate Professor, The Dartmouth Institute for Health Policy and Clinical Practice, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02000798
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: neurology; health communications
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIDEO (Experimental): Participants receive access to video recordings of their clinic visits
  Interventions: Other: HealthPAL
- Usual Care (No Intervention): Participants receive usual care (UC), which is their normal clinic visit and written after-visit summary

INTERVENTIONS:
Other: HealthPAL — Participants who are randomly assigned to the HealthPAL arm will have immediate post- visit access to audio/video-recordings of their clinical visit through a HIPAA-compliant web-based program called HealthPAL.
  Arms: VIDEO

SUMMARY:
Our objective in the proposed project is to: (a) operationalize and determine the feasibility and acceptability of a trial where clinic multi-disciplinary clinic (MDC) visits are audio/video recorded and shared with patients with ALS and their caregivers; (b) gather preliminary data examining the impact of routinely adding audio/video recordings of clinic visits to UC on self-management ability and other behavioral, health and health services outcomes at baseline (T0) and other regular interviews from enrollment (T1= 1 Week, T2= 3 Months); and (c) identify factors pertinent to the acceptability of our study protocol and the audio/video recording of visits.

DETAILED DESCRIPTION:
We will conduct a single-site, two-arm, parallel group, patient-randomized, controlled, pilot trial with 3-month follow up, to determine the feasibility, acceptability, and potential effectiveness of sharing audio/video recordings of multidisciplinary ALS clinics with patients and their caregivers. We will recruit 24 patients with ALS and their caregivers over a recruitment period of 1 year. We are primarily interested in determining the feasibility of the trial and acceptability of the audio/video intervention. We will also explore the impact on the patients' ability to self-manage their care as well as exploratory outcomes, at baseline (T0 = pre-visit), at T1 (1 week), and at T2 (3 months).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed and primarily treated for Amyotrophic Lateral Sclerosis (ALS)
* Aged 18 years or greater
* Can communicate in English (verbally, on a computer, or with assistance)
* Have email
* Have internet access
* Willing to have their multidisciplinary clinic visit audio/video recorded for a 3 month period

Exclusion Criteria:

* Those without the capacity to provide consent, either themselves or via proxy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Patient Enrollment (Feasibility) | Study Completion, an average of 1 year
  Meeting the targeted recruitment number and rate (two patients per month over a 12 month period)
Intervention Fidelity (Feasibility) | Three months
  The proportion of ALS MDC (multidisciplinary clinic) patients in the intervention arm that received the VIDEO intervention with full adherence to a pre-defined protocol fidelity checklist. Any deviations will be documented.
Patient use of the Intervention (Acceptability) | Three months
  The proportion of ALS MDC (multidisciplinary clinic) patients in the intervention arm who used the recording between the day of receipt and the three-month follow up

SECONDARY OUTCOMES:
Change from baseline in Patient Satisfaction, as measured by the Patient Satisfaction Questionnaire-18 (PSQ-18) | Baseline, one week, three months
  Scores are measured on an 18-item, 5-level scale, with a score of 1 indicating "strongly agree" and a score of 5 indicating "Strongly Disagree". Scores range from 18 to 90, with lower scores indicating higher levels of satisfaction.
Change from baseline in adherence to treatment, as measured by the Medical Outcomes Study - General Adherence | Baseline, one week, three months
  Scores are measured on a 5-item, 6-level scale, with a score of 1 indicating "None of the time" and a score of 6 indicating "All of the time". Scores range from 6 to 30, with higher scores indicating higher levels of adherence. Items 1 and 3 are scored in reverse.
Change from baseline in adherence to medications, as measured by the Adherence to Refills and Medications Scale - 7 (ARMS-7) | Baseline, one week, three months
  Scores are measured on a 7-item, 4-level scale, with a score of 1 indicating "None" and a score of 4 indicating "All". Scores range from 7 to 28, with lower scores indicating higher levels of adherence.
Change from baseline in adherence to physical therapy, as measured by the Exercise Adherence Rating Scale (EARS) | Baseline, one week, three months
  Scores are measured on a 6-item, 5-level scale, with 0 indicating "Completely agree" and 4 indicating "Completely disagree". Scores range from 0 to 30, where a higher score indicates a higher level of adherence.
Change from baseline in anxiety, as measured by the Generalized Anxiety Disorder - 7 (GAD-7) | Baseline, three months
  Scores are based on a 7-item, 4-level scale with 0 indicating "Not at all" and 3 indicating "Nearly every day". Higher scores indicate higher levels of anxiety.
Change from baseline in functional status, as measured by the Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) | Baseline, one week, three months
  Scores are measured on a 13-item, 5-level scale, with 0 indicating low function and 4 indicating high functioning, and one item as "yes/no". Scores range from 0 to 48, with high scores indicating higher levels of functioning.
Change from baseline in depression, as measured by the Patient Health Questionnaire - 8 (PHQ-8) | Baseline, three months
  Scores are based on a 8-item, 4-level scale with 0 indicating "Not at all" and 3 indicating "Nearly every day". Higher scores indicate higher levels of depression.
Level of Communication in the Visit, as measured by the Interpersonal Processes of Care (IPC) | One week
  Scores are based on an 18-item, 5-level scale with 1 indicating "Never" and 5 indicating "Always". Scores range from 18 to 90, with higher scores indicating higher levels of communication.
Level of literacy, as measured by the Single Item Literacy Screener | Baseline
  Scores are measured on a single item, 5-level scale. Scores range from 1 to 5, with higher scores indicating higher levels of literacy.
Change in caregiver burden, as measured by the Burden Scale for Family Caregivers - Short (BSFC-s) | Baseline, one week, three months
  Scores are based on a 10-item, 4-level scale, with 0 indicating strongly disagree and 3 indicating strongly agree. Scores range from 0 to 30, with higher scores indicate higher levels of burden.
Change in caregiver preparedness, as measured by the Preparedness for Caregiving Scale | Baseline, one week, three months
  Scores are based on a 9-item, 5-level scale, with 0 indicating not at all prepared, and 4 indicating very well prepared. Scores range from 0 to 45, with higher scores indicating higher levels of preparedness.
Change in self-efficacy, as measured by the Self Efficacy for Managing Chronic Disease scale | Baseline, one week, three months
  Scores are measured on 6x 10-item scales. Scores range from 0 to 60, with higher scores indicating higher levels of self-efficacy.
Feasibility of the Intervention, as measured by the Feasibility of Intervention Metric (FIM) | Three months from baseline
  Scores are measured on a 4-item, 5-level scale, with a score of 1 indicating "completely disagree" and 5 indicating "completely agree". Scores range from 4 to 20, with higher scores indicating higher levels of feasibility.
Acceptability of the Intervention, as measured by the Acceptability of Intervention Metric (AIM) | Three months from baseline
  Scores are measured on a 4-item, 5-level scale, with a score of 1 indicating "completely disagree" and 5 indicating "completely agree". Scores range from 4 to 20, with higher scores indicating higher levels of acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cohen, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Paul J Barr, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bratches RWR, Cohen J, Carpenter-Song E, Mistler L, Barr PJ. The Feasibility and Acceptability of Sharing Video Recordings of Amyotrophic Lateral Sclerosis Clinical Encounters With Patients and Their Caregivers: Pilot Randomized Clinical Trial. JMIR Form Res. 2024 Jun 26;8:e57519. doi: 10.2196/57519. PMID 38924779